CLINICAL TRIAL: NCT07320131
Title: Perceived Barriers and Facilitators to Physical Activity and Associated Factors Among Turkish Youth: A Cross-Sectional Study
Brief Title: Perceived Barriers and Facilitators to Physical Activity in Turkish Youth
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Assistant Professor, Istinye University
Other Study IDs: 1000
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Youth; Physical Activity; Barriers; Facilitators; Sleepiness
MeSH Terms: conditions — Motor Activity; Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth with aged 15-24

SUMMARY:
Physical activity is a key determinant of physical and mental health among youth; however, participation levels are often influenced by various perceived barriers and facilitators. Understanding these perceptions, together with related psychosocial factors, will provide valuable insights for the development of targeted interventions. This study will aim to investigate perceived barriers and facilitators to physical activity among Turkish youth and to examine their associations with physical activity levels, perceived stress, and daytime sleepiness. This cross-sectional study will include individuals aged 15-24 years. Participants' sociodemographic characteristics will be recorded. Data will be collected using four validated questionnaires administered in a face-to-face setting. Perceived barriers and facilitators to physical activity will be assessed using the Barriers and Facilitators to Youth Physical Activity Questionnaire (BFYPA). Physical activity levels will be evaluated using the short form of the International Physical Activity Questionnaire (IPAQ-SF). Perceived stress levels will be measured using the Perceived Stress Scale (PSS), and daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS). Appropriate statistical analyses will be performed to examine relationships between study variables.

ELIGIBILITY:
Inclusion Criteria:

* Being between 15 and 24 years old
* Being a volunteer

Exclusion Criteria:

* Having a musculoskeletal problem that may alter physical activity habits
* Having a cardiovascular or respiratory problem
* Having diabetes mellitus
* Taking chronic medication
* Having a body mass index of 35 kg/m2 or higher
* Having any other condition that would prevent physical activity

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The Physiotherapy and Rehabilitation Application and Research Center of Istinye University
Sampling Method: Non-Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The Barriers and Facilitators to Youth Physical Activity Questionnaire | 1 day
  The Barriers and Facilitators to Youth Physical Activity Questionnaire (BFYPA) will be used to assess perceived barriers and facilitators to physical activity among youth. The questionnaire will evaluate multiple dimensions of physical activity-related barriers and facilitators through standardized self-report items, with higher scores indicating greater perceived influence of barriers or facilitators.
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | 1 day
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF) will be used to assess participants' physical activity levels over the previous seven days. Physical activity will be quantified in metabolic equivalent task minutes per week (MET-min/week) based on the frequency and duration of walking, moderate-intensity, and vigorous-intensity activities.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | 1 day
  The Perceived Stress Scale (PSS) will be used to evaluate the degree to which participants perceive situations in their daily lives as stressful. The scale will assess perceived stress levels through a standardized self-report format, with higher scores indicating greater perceived stress.
Epworth Sleepiness Scale (ESS) | 1 day
  The Epworth Sleepiness Scale (ESS) will be used to assess daytime sleepiness by evaluating the likelihood of dozing or falling asleep during common daily activities. Higher total scores will indicate greater levels of daytime sleepiness.